CLINICAL TRIAL: NCT01264107
Title: An Open Study to Evaluate the Sustained Effect in Patients Showing Virological Responses With Muscle-related Symptom of Chronic Hepatitis B Patients Who Received Clevudine
Status: Completed | Type: Observational
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Hee Won Yoo, Bukwang Pharm. Co. Ltd.
Other Study IDs: CLV-409
Record Dates: First submitted 2010-12-19; First posted 2010-12-21 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An Open Study to Evaluate the Sustained Effect in Patients Showing Virological Responses With Muscle-related Symptom of Chronic Hepatitis B Patients Who Received Clevudine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients is currently clevudine treatment.
2. Patients with HBV DNA < 300 cpoies/mL and ALT normal Showing Muscle-related Symptom Who received Clevudine
3. Patient who is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
2. Patient is pregnant or breast-feeding.
3. Patient has a significant gastrointestinal, renal, decompensated liver, bronchopulmonary, neurological, cardiac, oncologic(except HCC)or allergic disease.
4. Patient, in the opinion of the investigator, unsuitable for the study.
5. Showing Muscle-related Symptom who any other evidence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An Open Study to Evaluate the Sustained Effect in Patients Showing Virological Responses With Muscle-related Symptom of Chronic Hepatitis B Patients Who Received Clevudine
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sustained antiviral activity effect | at week 48

SECONDARY OUTCOMES:
The change of sAg | at week 48
Proportion of sAg loss | at week 48
The change of HBV DNA form the baseline | at week 48
  (log copies/mL)
Proportion of patients with ALT normalization | at week 48
Proportion of HBeAg loss/seroconversion | at week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Soon Koo Baik, Wonju, Kangwon-do 162 Ilsan-dong, Wonju, Kangwon-do, South Korea